CLINICAL TRIAL: NCT05651841
Title: REVErsing Airway Remodelling With Tezepelumab : a Protocol for a Double-blind Randomized Controlled Trial for Patients With Asthma
Brief Title: REVErsing Airway Remodelling With Tezepelumab
Acronym: REVERT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL22_0123
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Airway Remodelling, Asthmatic
Keywords: exacerbating asthma; Severe asthma; Airway Remodelling
MeSH Terms: conditions — Airway Remodeling; Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo / Tezepelumab (Experimental): After 6-months of treatment, patients initially receiving placebo will switch to Tezepelumab for an additional 6 months.
  For 6 months of treatment, six subcutaneous (injections in accessorized pre-filled syringes (APFS)) are performed every 4 weeks. Each subcutaneous injection corresponds to 210 mg of Tezepelumab or analogous placebo.
  Interventions: Drug: Tezepelumab; Other: placebo
- Tezepelumab / Tezepelumab (Experimental): After 6-months of treatment, patients receiving Tezepelumab will continue Tezepelumab for an additional 6 months. For 6 months of treatment, six subcutaneous (injections in accessorized pre-filled syringes (APFS)) are performed every 4 weeks.Each subcutaneous injection corresponds to 210 mg of Tezepelumab.
  Interventions: Drug: Tezepelumab
- Tezepelumab / Placebo (Experimental): After 6-months of treatment, patients receiving Tezepelumab will be switched to a placebo for an additional 6 months.
  For 6 months of treatment, six subcutaneous (injections in accessorized pre-filled syringes (APFS)) are performed every 4 weeks. Each subcutaneous injection corresponds to 210 mg of Tezepelumab or analogous placebo.
  Interventions: Drug: Tezepelumab; Other: placebo

INTERVENTIONS:
Drug: Tezepelumab — Tezepelumab is supplied as a sterile, single-use, preservation-free, clear, colourless to slightly yellow liquid for subcutaneous administration in accessorized pre-filled syringes (APFS).
  Injections will be performed by study staff (doctors or nurses) during face-to-face study visits in participating centres.
  Subcutaneous injections are performed in a different body-part following the suggested rotation diagram.
Other: placebo — APFS containing analogous placebo identical in appearance:
  Injections will be performed by study staff (doctors or nurses) during face-to-face study visits in participating centres.
  Subcutaneous injections are performed in a different body-part following the suggested rotation diagram.
  Arms: Placebo / Tezepelumab; Tezepelumab / Placebo

SUMMARY:
The aim of this protocol is to perform a first randomized controlled trial evaluating how Tezepelumab affects the bronchial morphology (and computed tomographic variables in general) of asthmatic patients. In parallel, the investigators also hope to reproduce clinical benefits and perform a transcriptomic study that will juxtapose changes in genetic expression with changes in bronchial morphology and inflammatory signatures. The general hypothesis is that tezepelumab treatment is capable of at least partially reversing bronchial remodelling as detected on computed-tomographic (CT) scans. The investigators also expect such reversal to occur within a unique physiological repair environment that will be reflected by transcriptomic profiles

DETAILED DESCRIPTION:
Tezepelumab is a human IgG2l monoclonal antibody (mAb) directed against TSLP. Double-blind, randomized controlled trials comparing Tezepelumab treatment against placebo demonstrate net positive benefits in asthma patients. Animal research currently indicates that blocking TSLP can prevent bronchial remodelling in murine models (Chen et al. 2013), but no such observations have been attempted in humans. Within this context, the aim of this protocol is to perform a first randomized controlled trial evaluating how Tezepelumab affects the bronchial morphology (and computed tomographic variables in general) of asthmatic patients. In parallel, the investigators also hope to reproduce clinical benefits and perform a transcriptomic study that will juxtapose changes in genetic expression with changes in bronchial morphology and inflammatory signatures.

The general hypothesis is that tezepelumab treatment is capable of at least partially reversing bronchial remodelling as detected on computed-tomographic (CT) scans. The investigators also expect such reversal to occur within a unique physiological repair environment that will be reflected by transcriptomic profiles.

The primary objective of this protocol is therefore to compare the change-from-baseline in the average percentage bronchial wall area (%WA = (wall area (mm2)/ (wall area (mm2) + lumen area (mm2)))×100) for patients with asthma and undergoing 6 months of tezepelumab treatment with a similar population treated via placebo. Secondarily, continued treatment effects associated with longer treatment (12 months) or remanence after treatment stopping at 6 months will also be quantified. Study arms will additionally be compared in terms of:

* Changes in radiomics (CT-scan data);
* Changes in exacerbation rates and lung function;
* Changes in serum club cell secretory protein (CCSP);
* Changes in nasal single-cell transcriptomic signatures.

This study also has an exploratory component designed to characterize the physiological repair environment. In depth radiomic and transcriptomic (including single-cell analyses) profiling will be performed. Finally, the capacity of baseline data to predict the response to tezepelumab will also be explored.

ELIGIBILITY:
Inclusion Criteria:

Admitted to screening visit:

* Minimum age: 18
* Maximum age: 85
* Able to perform an inspiratory and expiratory thoracic computed tomography (CT) scan, plus a nasal CT
* In stable condition for CT scan
* Physician-diagnosed asthma according to GINA criteria
* Disease with clinical impact: at least 1 severe or 2 moderate exacerbations in the previous 12 months despite treatment according to the best standards of care
* Maximal inhaled therapy comprising high dose ICS and at least a second controller according to GINA

Based on results of screening visit and run-in:

* Post-bronchodilator forced expiratory volume in 1 second (FEV1) predicted values must be at 25-90%
* Asthma Control Questionnaire 6 (ACQ6) > 1.5
* Oral corticosteroid maintenance therapy (if used) ≤7.5 mg/day
* On CT scan, the average percentage wall area index at the B1 and B8 bronchi (generation 3, 4, 5) is >65%

Exclusion Criteria:

* CT abnormalities evocative of any respiratory condition other than asthma
* Treatment regimen discordant with best practices
* Pulmonary disease other than asthma requiring treatment during the previous 12 months
* A smoking history of >20 pack years
* Receipt of any marketed or investigational biologic agent§ within 3 months or 5 halflives (whichever is longer) prior to randomization or receipt of any investigational non biologic agent within 30 days or 5 half-lives (whichever is longest) prior to randomization or receipt of live attenuated vaccines 30 days prior to the date of randomization. Participants enrolled in current or previous tezepelumab studies will not be included. Participants on previous biologics treatment are allowed to enter the study provided the appropriate washout period is fulfilled.
* Absence of signed consent
* Non-beneficiary of the French social security, single-payer health insurance system
* Presence of any condition (physical, psychological or other) that might, in the investigator's opinion, hinder study performance
* The patient is unavailable or unwilling to participate in future visits
* Potential interference from other studies
* Protected populations according to the French public health code
* Male or female patients seeking to conceive a child
* Women of childbearing potential and fertile men not using birth control method
* Pregnant, breastfeeding or lactating women
* History of a clinically significant infection, including upper (URTI) or lower respiratory tract infection (LRTI), requiring treatment with antibiotics or antiviral medications finalised < 2 weeks before randomization. Patients with preexisting serious infections should be treated before initiating therapy with tezepelumab.
* A helminth parasitic infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
* Patients using vaping products, including electronic cigarettes (because may induce abnormality at CT scan).
* Bronchial thermoplasty in the last 12 months prior to Visit 1.
* History of documented immune complex disease (Type III hypersensitivity reactions) following any biologic therapy.
* History of known immunodeficiency disorder including a positive human immunodeficiency virus test or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
* Receipt of the T2 cytokine inhibitor Suplatast tosilate within 15 days prior to randomization.
* Treatment with systemic immunosuppressive/immunomodulating drugs (eg, methotrexate, cyclosporine, etc.), except for OCS used in the treatment of asthma/asthma exacerbations, within the last 12 weeks or 5 half-lives (whichever is longer) prior to randomization.
* Receipt of immunoglobulin or blood products within 30 days prior to randomization.
* Receipt of allergen immunotherapy not stable within 30 days prior to randomization or with anticipated change during the treatment period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparaison on CT-scan in the change in mean percentage bronchial wall area (%WA) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  %WA = (wall area (mm²)/ (wall area (mm²) + lumen area (mm²)))×100) at bronchial levels likely to be affected.

SECONDARY OUTCOMES:
compare on CT-scan the change in mean %WA between arms | Between baseline and 12 months
  %WA = (wall area (mm2)/ (wall area (mm2) + lumen area (mm2)))×100) at bronchial levels likely to be affected.
Comparaison on CT-scan in the average percentage bronchia wall thickness index (%WT) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  %WT = (wall thickness (mm) / airway diameter (mm))×100
Comparaison on CT-scan in the average percentage bronchia wall thickness index (%WT) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 12 months
  %WT = (wall thickness (mm) / airway diameter (mm))×100
compare on CT-scan the change in wall area at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  lumen area (mm²)
compare on CT-scan the change in lumen area at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  lumen area (mm²)
compare on CT-scan the change in ratio wall area (WA) / lumen area(LM) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  WA/LA = WA(mm²)/LA(mm²)
compare on CT-scan the change in lumen diameter at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  lumen diameter (mm)
compare on CT-scan the change in lumen circularity at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  lumen circularity (4pi x area x perimeter-²)
Comparaison on CT-scan in the average percentage bronchial wall area(%WA) corrected by body surface area(BSA) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  %WA/BSA = (wall area (mm²)/ (wall area (mm²) + lumen area (mm²))×100)/(0.007184 x weight (kg)^0.425 x height (cm) ^0.725)
Comparaison on CT-scan in the average percentage bronchial wall thickness (%WT) corrected by body surface area(BSA) at the B1 and B8 bronchi, generations 3, 4 and 5 | Between baseline and 6 months
  %WT/BSA = ((wall thickness (mm) / airway diameter (mm))×100)/(0.007184 x weight (kg)^0.425 x height (cm) ^0.725)
Change in the expiratory to inspiration ratio of mean lung density (MLDe/i), | At Baseline, 6 months and 12 months
  expiratory-to-inspiratory ratios of mean lung density (MLDe/i)
Quantitative computed tomography measurements to evaluate airflow obstruction | At Baseline, 6 months and 12 months
  Mucus plugging score (MPS)
Change in Total small Airway Count (TAC) | Between Baseline and 6 months
  Total small Airway Count (TAC) mesured with Quantitative computed tomography
Change in Total small Airway Count (TAC) | Between Baseline and 12 months
  Total small Airway Count (TAC) mesured with Quantitative computed tomography
Change in Lund Mackay score | Between Baseline and 6 months
  Each sinus group (maxillary, anterior ethmoids, posterior ethmoids, sphenoid, frontal, ostiomeatal complex) is graded between 0 and 2 (0: no abnormality; 1: partial opacification; 2: total opacification). The ostiomeatal complex is scored as "0" (not obstructed) or "2" (obstructed). A total score of 0-24 is possible, and each side can be considered separately (0-12)
Change in Lund Mackay score | Between Baseline and 12 months
  Each sinus group (maxillary, anterior ethmoids, posterior ethmoids, sphenoid, frontal, ostiomeatal complex) is graded between 0 and 2 (0: no abnormality; 1: partial opacification; 2: total opacification). The ostiomeatal complex is scored as "0" (not obstructed) or "2" (obstructed). A total score of 0-24 is possible, and each side can be considered separately (0-12)
Change in Presence/absence of nasal polyposis | Between Baseline and 6 months
  Nasal brushing
Change in Presence/absence of nasal polyposis | Between Baseline and 12 months
  Nasal brushing
Change in Annualized exacerbation rates | Between Baseline and 12 months
  The patient journal will cover exacerbations and hospitalizations.Exacerbations will be further characterized according to severity as defined by GINA. Episode data (hospitalizations, and exacerbations) will be characterized by their beginning and end dates; These data will be used to estimate annualized exacerbation rates.
Change in Days alive and not exacerbating | Between Baseline and 12 months
  The patient journal will cover exacerbations and hospitalizations. Exacerbations will be further characterized according to severity as defined by GINA. Episode data (hospitalizations, and exacerbations) will be characterized by their beginning and end dates; These data will be used to estimate days alive and not exacerbating.
Change in Days alive and not hospitalized | Between Baseline and 12 months
  The patient journal will cover exacerbations and hospitalizations. Episode data (hospitalizations, and exacerbations) will be characterized by their beginning and end dates; These data will be used to estimate days alive and not hospitalized (total, and for each GINA type of exacerbation).
Change in forced expiratory volume in 1 second | Between Baseline and 6 months
  Pre- and post-bronchodilator spirometry (FEV1; litres and percent predicted)
Change in forced expiratory volume in 1 second | Between Baseline and 12 months
  Pre- and post-bronchodilator spirometry (FEV1; litres and percent predicted)
Change in forced vital capacity | Between Baseline and 6 months
  Pre- and post-bronchodilator spirometry (FVC; litres and percent predicted)
Change in forced vital capacity | Between Baseline and 12 months
  Pre- and post-bronchodilator spirometry (FVC; litres and percent predicted)
Change in forced expiratory volume in 1 second / forced vital capacity Ratio | Between Baseline and 6 months
  Pre- and post-bronchodilator spirometry ( FEV1/FVC ratio (litres/litres)))
Change in forced expiratory volume in 1 second / forced vital capacity Ratio | Between Baseline and 12 months
  Pre- and post-bronchodilator spirometry ( FEV1/FVC ratio (litres/litres)))
Change in total lung capacity | Between Baseline and 6 months
  Pre-bronchodilator plethysmography (TLC(total lung capacity ); litres and percent predicted)
Change in total lung capacity | Between Baseline and 12 months
  Pre-bronchodilator plethysmography (TLC(total lung capacity ); litres and percent predicted)
Change in residual volume | Between Baseline and 6 months
  Pre-bronchodilator plethysmography (RV (residual volume ); litres and percent predicted)
Change in residual volume | Between Baseline and 12 months
  Pre-bronchodilator plethysmography (RV (residual volume ); litres and percent predicted)
Change in total lung capacity (TLC)/ residual volume(RV) ratio | Between Baseline and 6 months
  Pre-bronchodilator plethysmography : total lung capacity (TLC)/ residual volume(RV) ratio (litres/litres)
Change in total lung capacity (TLC)/ residual volume(RV) ratio | Between Baseline and 12 months
  Pre-bronchodilator plethysmography : total lung capacity (TLC)/ residual volume(RV) ratio (litres/litres)
Change in mean ACQ (Asthma Control Questionnaire)-6 score | Between Baseline and 6 months
  The ACQ6 is a shortened version of the ACQ((Asthma Control Questionnaire) that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score.
  Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions.
  Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma (Juniper et al. 2006). Individual changes of at least 0.5 are considered to be clinically meaningful.
Change in mean ACQ (Asthma Control Questionnaire)-6 score | Between Baseline and 12 months
  The ACQ6 is a shortened version of the ACQ((Asthma Control Questionnaire) that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and SABA use) omitting the FEV1 measurement from the original ACQ score.
  Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions.
  Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma (Juniper et al. 2006). Individual changes of at least 0.5 are considered to be clinically meaningful.
Change in Breathlessness, Cough and Sputum Scale (BCSS) | Between Baseline and 6 months
  The Breathlessness, Cough and Sputum Scale (BCSS) has undergone a vigorous validation process and is designed to assess patients' daily respiratory symptoms. Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms. A mean change in BCSS total score > 1.0 represents substantial symptomatic improvement, changes of approximately 0.6 can be interpreted as moderate, and changes of 0.3 can be considered small (DeVries et al. 2016; Leidy et al. 2003).
Change in Breathlessness, Cough and Sputum Scale (BCSS) | Between Baseline and 12 months
  The Breathlessness, Cough and Sputum Scale (BCSS) has undergone a vigorous validation process and is designed to assess patients' daily respiratory symptoms. Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms. A mean change in BCSS total score > 1.0 represents substantial symptomatic improvement, changes of approximately 0.6 can be interpreted as moderate, and changes of 0.3 can be considered small (DeVries et al. 2016; Leidy et al. 2003).
Change in Sino Nasal Outcome Test 22 | Between Baseline and 6 months
  The SNOT-22 is a further modification of the SNOT-20 (Piccirillo et al. 2002), where the scoring has been simplified by removing the importance rating. In addition to the normal 20-item version of the SNOT, 2 additional items were measured, nasal blockage, and loss of sense of taste and smell. The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes); a MCID of 8.90 has been established.
Change in Sino Nasal Outcome Test 22 | Between Baseline and 12 months
  The SNOT-22 is a further modification of the SNOT-20 (Piccirillo et al. 2002), where the scoring has been simplified by removing the importance rating. In addition to the normal 20-item version of the SNOT, 2 additional items were measured, nasal blockage, and loss of sense of taste and smell. The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes); a MCID of 8.90 has been established.
Change in St George Respiratory Questionnaire (SGRQ) | Between Baseline and 6 months
  The SGRQ is a 50-item patient-reported instrument developed to measure the health status of patients with obstructive airway diseases. The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition.
  The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
Change in St George Respiratory Questionnaire (SGRQ) | Between Baseline and 12 months
  The SGRQ is a 50-item patient-reported instrument developed to measure the health status of patients with obstructive airway diseases. The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition.
  The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
Change in ECRHS III Main Questionnaire | Between Baseline and 6 months
  The European Community Respiratory Health Survey (ECRHS) III Main questionnaire is a survey used to track changing respiratory situations within the general population for epidemiological purposes. The questionnaire is composed of 32 pages and 105 questions. For the purposes of the present study, only the questions 21-28 will be used. Each selected question will be used as a stand-alone variable.
  The advantage of using these questions is that study distributions and longitudinal change in results can be compared to previously published epidemiological results for the general population
Change in ECRHS III Main Questionnaire | Between Baseline and 12 months
  The European Community Respiratory Health Survey (ECRHS) III Main questionnaire is a survey used to track changing respiratory situations within the general population for epidemiological purposes. The questionnaire is composed of 32 pages and 105 questions. For the purposes of the present study, only the questions 21-28 will be used. Each selected question will be used as a stand-alone variable.
  The advantage of using these questions is that study distributions and longitudinal change in results can be compared to previously published epidemiological results for the general population
Changes in serum Club cell secretory protein (CCSP) | Between baseline and 6 months
  Changes in serum Club cell secretory protein (CCSP), an emerging blood marker associated with pulmonary function and cellular cross-talk
Changes in serum Club cell secretory protein (CCSP) | Between baseline and 12 months
  Changes in serum Club cell secretory protein (CCSP), an emerging blood marker associated with pulmonary function and cellular cross-talk
Number of adverse event between arms | Between baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU Dijon, Dijon
  - CHU Grenoble Alpes La Tronche, Grenoble
  - APHP Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Nord Marseille, Marseille
  - CHU de Montpelier, Montpellier
  - APHP Bichat, Paris
  - Hôpital Foch, Paris
  - Hôpital Haut-Lévêque, Pessac
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided